CLINICAL TRIAL: NCT05824299
Title: Influence of General Anesthesia Versus Spinal Anesthesia on Circulating Tumor Cells in Patients Undergoing Transurethral Resection of Bladder Tumor
Brief Title: Influence of Anesthesia Methods on CTCs in TURBT Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jie Tian, Principal Investigator, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CTC20230408
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Bladder Cancer
Keywords: Circulating Tumor Cells; General Anesthesia; Spinal Anesthesia; Transurethral Resection of Bladder Tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplastic Cells, Circulating | interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (Active Comparator): Patients in this group will receive general anesthesia during TURBT.
  Interventions: Procedure: General Anesthesia
- Spinal Anesthesia (Experimental): Patients in this group will receive spinal anesthesia during TURBT.
  Interventions: Procedure: Spinal Anesthesia

INTERVENTIONS:
Procedure: General Anesthesia — Patients will have TURBT under general anesthesia, which is induced with midazolam, propofol, sufentanil and rocuronium. The patients will be mechanically ventilated with laryngeal mask airway (LMA). Anesthesia will be maintained with sevoflurane/desflurane, propofol and remifentanil.
  Arms: General Anesthesia
Procedure: Spinal Anesthesia — Patients will have TURBT under spinal anesthesia. 10~15mg of 0.5% ropivacaine will be injected in the subarachnoid cerebrospinal fluid at the levels of L2-L3 or L3-L4 in lumbar space. It will numb the nerve supply of the belly, hips, bottom as well as legs. The patient stays awake and won't feel any pain due to operation.
  Arms: Spinal Anesthesia

SUMMARY:
Multiple lines of evidence have shown that anesthesia method is associated with long-term outcomes in patients undergoing surgery due to cancers, including lung, breast, prostate, and bladder cancer, etc. Circulating tumor cells (CTCs) have been validated as prognostic biomarkers of a number of cancers. The aim of this study is to investigate the effects of anesthesia methods on the number of CTCs in patients receiving transurethral resection of bladder tumor (TURBT). The difference of anesthesia method is achieved by using general anesthesia in one group and spinal anesthesia in the other group.

ELIGIBILITY:
Inclusion Criteria:

1. .≤18 Age ≤85，ASAI-III.
2. .Patients with primary bladder cancer of Stage T1 to T4, who are scheduled for transurethral resection of bladder tumor.
3. .Written informed consent.

Exclusion Criteria:

1. History of surgery within 6 months.
2. Contraindications for spinal anesthesia.
3. With a history of any other malignancy.
4. Having received preoperative neoadjuvant therapy.
5. History of long-term opioid use.
6. Combined with autoimmune diseases or having a history of prolonged hormone use or immunosuppressant use within 1 year.
7. Combined with impaired liver function (Child - Pugh C) or renal insufficiency (serum creatinine level over 442μmol•L-1).
8. Known hypersensitivity or suspected allergy to intervention drugs.
9. Proposed postoperative admission to ICU.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the number of Circulating Tumor Cells | on the Day 7~10 after surgery
  The number of circulating tumor cells will be measured by collecting 5 ml of venous blood sample.

SECONDARY OUTCOMES:
Surgeon Satisfaction | immediately after surgery
  The surgeon satisfaction will be measured with the Likert scale, which ranges from 0 to 50, with a higher score indicating higher satisfaction.
Patient Satisfaction | within 24 hours after surgery
  The patient satisfaction will be measured with the Modified Bauer Scale, which ranges from 0 to 50, with a higher score indicating higher satisfaction.
Visual Analogue Scale | at 24 hours after surgery
  Pain intensity will be assessed using the Visual Analogue Scale, which ranges from 0 to 10, with a higher score indicating greater pain intensity at 24 hours after surgery.
Nausea Score | at 24 hours after surgery
  Nausea score will be assessed using the Numerical Rating Scale, which ranges from 0 to 10, with a higher score indicating greater nausea ou score at 24 hours after surgery.
Hospitalization Days | up to 30 days
  The length of hospital stay will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital affliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No